CLINICAL TRIAL: NCT00821574
Title: Project to Promote the Evaluation of the Cardiovascular Risk in the Clinical Practice and to Evaluate Its Evolution Following the Implementation of a Preventive Multifactorial Strategy Aimed to Reduce the Total Risk Level (SCORE Algorithm), in Subjects Suffering From Metabolic Syndrome and With a Risk Level ≥5%
Brief Title: Reducing the Overall Risk Level in Patients Suffering From Metabolic Syndrome
Acronym: LesScore
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CXUO320BIT02
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Hypertension, Dyslypidaemia
Keywords: Hypertension, dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — Fluvastatin; Valsartan; Hydrochlorothiazide

ARMS (3):
- 1 (Experimental): Fluvastatin: daily 80 mg, oral
  Interventions: Drug: Fluvastatin
- 2 (Experimental): Valsartan
  Interventions: Drug: Valsartan
- 3 (Experimental): Hydrochlorothiazide
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Fluvastatin — Fluvastatin: daily 80 mg, oral
  Other Names: Lescol
  Arms: 1
Drug: Valsartan — Valsartan: daily 160 mg, oral
  Other Names: Diovan
  Arms: 2
Drug: Hydrochlorothiazide — Hydrochlorothiazide: daily 12.5mg, oral
  Arms: 3

SUMMARY:
This study will evaluate the efficacy of a multi factorial preventive scheme of action (including fluvastatin and valsartan) to reduce the overall risk level in patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 - 65 years
* Diagnosed metabolic syndrome
* Risk of cardiovascular death ≥ 5% (according to SCORE)
* Written informed consent

Exclusion Criteria:

* Women not in menopause or not using efficient contraception
* Known hypersensitivity to study drugs
* History of ischemic heart disease

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2005-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Change in global risk from baseline to 3 and 9 months, as evaluated by the SCORE algorithm | 9 months

SECONDARY OUTCOMES:
Change from baseline after 3 and 9 months in the individual risk factors (e.g. blood pressure, lipid variables) | 9 month
Proportion of patients with controlled glycemia | 9 months
Percentage of patients no longer classifiable as having metabolic syndrome | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Rossi, MD, Principal Investigator — ASL Terni 4, Narni (TR) - Italy

REFERENCES:
- [Result] Ambrosioni E, Cicero AF, Parretti D, Filippi A, Rossi A, Peruzzi E, Borghi C. Global cardiovascular disease risk management in italian patients with metabolic syndrome in the clinical practice setting. High Blood Press Cardiovasc Prev. 2008 Apr;15(2):37-45. doi: 10.2165/00151642-200815020-00001. Epub 2013 Jan 3. PMID 23334870